CLINICAL TRIAL: NCT00418717
Title: An Open-label, Multicenter, Dose-regimen Study Evaluating the Efficacy and Safety of Etanercept 50 mg Once-weekly Dose in Japanese Subjects With Rheumatoid Arthritis
Brief Title: Open Label, Dose-Regimen Study Evaluating Etanercept 50 mg Once-Weekly In Japanese Subjects With RA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-321
Record Dates: First submitted 2007-01-02; First posted 2007-01-05 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Arm 1: Period A-25mg BW; Arm 1: Period B-50mg QW
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Period A: Weeks 1-4: Etanercept 25mg (25mg vial)bi-weekly (BW); Period B: Weeks 5-12: Etanercept 50mg (50mg vial) weekly (QW)

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of a once-weekly dose of etanercept for rheumatoid arthritis. Currently, patients in Japan can only use 25 mg etanercept two times a week. If a once-a-week regimen of 50 mg is approved, this would be more convenient for most patients. This once-weekly regimen is used in countries outside of Japan.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects of Japanese ancestry and living in Japan.
* Subjects who are receiving the approved dose of 25 mg etanercept BIW for at least 6 months and have stable disease activity, as determined by investigator's judgment for 3 months before test articles administration.
* Subjects who have mildly active rheumatoid arthritis as demonstrated by 5 swollen joints and 5 tender/painful joints.

Main Exclusion Criteria:

* Prior treatment with Disease Modifying Anti-Rheumatic Drugs (DMARDs) and/or methotrexate (MTX) within 6 months of the baseline visit.
* Subjects considered being in disease remission, per investigator's judgment.
* Received other biological drugs, rituximab, anti-CD-4 agents, or diphtheria interleukin-2 fusion protein (DAB-IL-2) within 6 months prior to baseline.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (12):
- Japan (12):
  - Nunoya-cho Goshogawara, Aomori
  - Kokubu, Kurume, Fukuoka
  - Inomachi Takasaki, Gunma
  - Higashiuneno Kawanishi, Hyōgo
  - Mukogawa-cho, Nishinomiya, Hyōgo
  - Kamiyokoba, Tsukuba, Ibaraki
  - Douhaku, Suzuka, Mie-ken
  - Hazama, Isobe-cho, Shima, Mie-ken
  - Hisai Myojin-cho, Tsu, Mie-ken
  - Yamato, Sasebo, Nagasaki
  - Higashizuka, Kurashiki, Okayama-ken
  - Toranomon, Minato-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Japan from January 2007 to September 2007.
Pre-assignment Details: Subjects were screened up to 4 weeks and received 25 mg etanercept (as test article) BW for 4 weeks during treatment period A. At the end of the period A, the same cohort of subjects entered period B and received etanercept 50 mg (as test article) QW for 8 weeks to assess the efficacy and safety of a QW regimen.
Groups:
- Etanercept (ETN): Weeks 1-4 (Treatment period A): Etanercept 25 mg bi-weekly (BW)
  Weeks 5-12 (Treatment period B): Etanercept 50mg once weekly (QW)
Period: Treatment Period A - Weeks 1-4
Arm/Group | Etanercept (ETN)
Started | 42
Completed | 41
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Treatment Period B - Weeks 5-12
Arm/Group | Etanercept (ETN)
Started | 41
Completed | 39
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 53.14 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score Using 28-joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4ESR) by Treatment Period.
Description: DAS28-4ESR is a clinical index of rheumatoid arthritis disease activity based on information from swollen joints, tender joints, acute phase response (Erythrocyte Sedimentation Rate) and general health. DAS28-4ESR scores range from 0 - 10, where a score of less than or equal to 3.2 implies well controlled disease and greater than or equal to 5.1 implies active disease. In this analysis, the DAS28-4ESR is compared for 2 different treatment regimens (used sequentially by the same patient population): Treatment Period A: ETN 25 mg BW (at week 4) vs Treatment Period B: ETN 50 mg QW (at week 12).
Time Frame: weeks 4 and 12
Population: The analysis population was modified intent to treat (mITT), which included all patients who completed the 25 mg BW dose treatment period and received at least 1 dose of 50 mg OW. Data on observed cases: 41 patients from ENT 25 mg BW (week 4) and 39 patients from ETN 50 mg OW (week 12).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 39
units on scale
  Treatment Period A: ETN 25mg BW (week 4) | 3.26 (0.66)
  Treatment Period B: ETN 50mg QW (week 12) | 3.13 (0.65)
Statistical Analysis 1: Comparison: Etanercept (ETN); Test type: Superiority or Other; Mean Difference (Net) = -0.10, 95% CI [-0.25 to 0.06]

2. Secondary Outcome: Area Under the Concentration-Time Curve (AUC)
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. In this analysis, the AUC is compared for 2 different treatment regimens (used sequentially by the same patient population): Treatment Period A: ETN 25 mg BW (at week 4) vs Treatment Period B: ETN 50 mg QW (at week 12). Blood samples were taken on day 0 of PK analysis and collected every day after for 7 days for weeks 4 and 12.
Time Frame: 7 days after week 4 and 7 days after week 12
Population: The analysis population was the Pharmacokinetic (PK) subset, which included all patients who completed the 25 mg BW dose treatment period, received at least 1 dose of 50 mg QW and elected to participate in the PK assessment. Data on observed cases: 18 patients from ETN 25 mg BW (week 4) and 17 patients from ETN 50 mg QW (week 12).
Measure: Mean (Standard Deviation); unit: ug*Day/mL
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 17
ug*Day/mL
  Treatment Period A: ETN 25mg BW (week 4) | 19.67 (5.7)
  Treatment Period B: ETN 50mg QW (week 12) | 17.92 (6.09)

ADVERSE EVENTS:
Arm/Group | Etanercept (ETN)
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Etanercept (ETN)
Calculus Ureteric / Pyelonephritis (Renal and urinary disorders) | 1/41
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Etanercept (ETN)
Abdominal pain (Gastrointestinal disorders) | 1/42
Abdominal pain upper (Gastrointestinal disorders) | 1/42
Infections and Infestations (Infections and infestations) | 12/42
Dry mouth (Gastrointestinal disorders) | 1/42
Gastric ulcer (Gastrointestinal disorders) | 1/42
Gingivitis (Gastrointestinal disorders) | 1/42
Parotid gland enlargement (Gastrointestinal disorders) | 1/42
Stomatitis (Gastrointestinal disorders) | 2/42
Tongue ulceration (Gastrointestinal disorders) | 1/42
Toothache (Gastrointestinal disorders) | 1/42
Vomiting (Gastrointestinal disorders) | 1/42
Chest pain (General disorders) | 1/42
Odema peripheral (General disorders) | 1/42
White blood cell count increase (Investigations) | 1/42
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/42
Dizziness (Nervous system disorders) | 3/42
Headache (Nervous system disorders) | 2/42
Calculus ureteric (Renal and urinary disorders) | 1/42
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/42
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1/42
Ecchymosis (Skin and subcutaneous tissue disorders) | 1/42
Photodermatosis (Skin and subcutaneous tissue disorders) | 1/42
Rash (Skin and subcutaneous tissue disorders) | 1/42
Hypertension (Vascular disorders) | 2/42
Pyrexia (General disorders) | 1/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.